CLINICAL TRIAL: NCT00747305
Title: Biomarkers of Tumor Angiogenesis and Response to Sunitinib Maleate in Renal Cell Carcinoma
Brief Title: Sunitinib Before and After Surgery in Treating Patients With Metastatic Kidney Cancer That Can Be Removed By Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated early due to low accrual.
Sponsor: Harry Drabkin (Other)
Responsible Party: Sponsor-Investigator, Harry Drabkin, Director, Hematology Oncology Division, Medical University of South Carolina
Organization: Medical University of South Carolina (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000612590; MUSC-101219
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-04

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; clear cell renal cell carcinoma; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Sunitinib; Gene Expression Profiling; Reverse Transcriptase Polymerase Chain Reaction; Blotting, Western; Immunohistochemistry; Chemotherapy, Adjuvant; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sunitinib (Experimental): Sunitinib will be administered for 8 weeks prior to sugery
  Interventions: Drug: sunitinib malate; Genetic: gene expression analysis; Genetic: reverse transcriptase-polymerase chain reaction; Genetic: western blotting; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Procedure: adjuvant therapy; Procedure: neoadjuvant therapy; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: sunitinib malate
Genetic: gene expression analysis
Genetic: reverse transcriptase-polymerase chain reaction
Genetic: western blotting
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Procedure: adjuvant therapy
Procedure: neoadjuvant therapy
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving sunitinib before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving it after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This clinical trial is studying how well sunitinib works when given before and after surgery in treating patients with metastatic kidney cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* To describe the gene expression of VEGF and non-VEGF angiogenic growth factor genes in kidney cancer specimens from patients with metastatic renal cell carcinoma treated with sunitinib malate.
* To describe the association between quantitative gene expression levels of VEGF and non-VEGF angiogenic factors and clinical efficacy of this drug, as measured by response, duration of response, and time to progression in these patients.

OUTLINE: Patients receive oral sunitinib malate once daily for 8 weeks. Within 2 weeks after completion of neoadjuvant chemotherapy, patients undergo a nephrectomy and evaluation for response to therapy. Beginning 4-8 weeks after surgery patients resume oral sunitinib malate once daily for up to 12 months in the absence of disease progression or unacceptable toxicity.

Patients with disease progression after 8 weeks of adjuvant treatment receive treatment off study with other agents.

Viable (non-necrotic) tumor and non-tumor kidney tissue samples are obtained at the time of nephrectomy for correlative biomarker studies. Tissue samples are analyzed for gene expression of VEGF and non-VEGF angiogenic factors by real-time RT-PCR, western blot, and/or IHC. Blood samples are obtained at baseline and at 4 and 8 weeks for evaluation of circulating levels of VEGF and selected chemokines.

After completion of study therapy, patients are followed monthly.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of clear cell renal cell carcinoma

  * Metastatic disease
  * Primary tumor is considered amenable to surgery
* Measurable disease, defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension (longest diameter to be recorded) as > 20 mm by conventional techniques or as > 10 mm by spiral CT scan
* No untreated brain metastases

  * Treated brain metastases allowed provided lesion has been stable on two consecutive CT or MRI scans separated by ≥ 2 months

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Leukocytes ≥ 3,000/μL
* ANC ≥ 1,500/μL
* Platelet count ≥ 75,000/μL
* Hemoglobin ≥ 8.5 g/dL
* Total Bilirubin ≤ 2 times upper limits of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Creatinine ≤ 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to undergo nephrectomy and treatment with sunitinib malate
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to sunitinib malate
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements

PRIOR CONCURRENT THERAPY:

* No prior systemic treatment with sunitinib malate
* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients
* Concurrent medications or substances known to affect, or with the potential to affect, the activity or pharmacokinetics of sunitinib malate allowed at the discretion of the principal investigator

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Describe the gene expression of VEGF and non-VEGF from eligible patients being treatment with Sunitinib. | at various points throughout the study duration
Describe the association between quantitative gene expression levels of VEGF and non-VEGF angiogenic factors with the clinical efficacy of Sunitinib as measured by response, duration or response and time to progression | at various points throughout the study duration

CONTACTS AND LOCATIONS:
Overall Officials: Harry A. Drabkin, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina, United States